CLINICAL TRIAL: NCT05365685
Title: Effect of the Degree of Energy Turnover on Appetitive Responses in Adolescents With Obesity
Brief Title: Energy Turnover and Appetite
Acronym: NEXT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RBHP 2021 BOIRIE 2; 2021-A02867-34 (Other: Clermont Ferrand University Hospital)
Record Dates: First submitted 2022-03-29; First posted 2022-05-09 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2022-03

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adolescents with obesity (Experimental): There is only one arm as this is an acute randomized study comparing three different conditions within the same sample of participants.
  Interventions: Behavioral: Low energy turnover

INTERVENTIONS:
Behavioral: Low energy turnover — Low Energy Turnover. The adolescents with ingest low energy intake at lunch and breakfast and will not perform physical exercise during the day. The will will receive an ad libitum meal at dinner time. Their food reward will be assessed before dinner. Their appetite feelings will be assessed at regular intervals.
  Moderate Energy Turnover. The adolescents with ingest moderate energy intake at lunch and breakfast and will perform one 45 minutes physical exercise during the day. The will will receive an ad libitum meal at dinner time. Their food reward will be assessed before dinner. Their appetite feelings will be assessed at regular intervals.
  High Energy Turnover. The adolescents with ingest high energy intake at lunch and breakfast and will perform two 45-minute physical exercises during the day. The will will receive an ad libitum meal at dinner time. Their food reward will be assessed before dinner. Their appetite feelings will be assessed at regular intervals.
  Other Names: Moderate energy turnover; High energy turnover

SUMMARY:
The aim of the study is to compare the effect of a low versus moderate versus high energy turnover on energy intake, appetite and food reward, in adolescents with obesity. 18 adolescents with obesity will then complete three experimental sessions in a randomized order: low, high and moderate Energy turnover.

DETAILED DESCRIPTION:
A total of 18 adolescents with obesity, aged 12-16 years olds will complete three experimental sessions in a randomized order: i) low energy turnover; ii) Moderate energy turnover and ; iii) High energy turnover. Their ad libitum energy intake at dinner will be assessed through an ad libitum buffet-type meal, their food reward assessed right before the dinner meal and their appetite sensation at regular intervals during the day.

ELIGIBILITY:
Inclusion Criteria:

* BMI percentile > 97th percentile according to the french curves.
* ages 12-16 years old
* Signed consent form
* being registered in the national social security system
* no contraindication to physical activity

Exclusion Criteria:

Previous surgical interventions that is considered as non-compatible with the study.

* Diabetes
* weight loss during the last 6 months
* cardiovascular disease or risks

Ages: 12 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2022-08-27 (Actual); Primary Completion 2022-10-29 (Actual); Study Completion 2023-11-08 (Actual)

PRIMARY OUTCOMES:
Energy intake measured during an ad libitum buffet meal (in kcal). | it will be assessed at dinner baseline
  food intake will be measured ad libitum during a dinner buffet. The adolescents will be offered an ad libitum buffet-type meal composed based on their food intake preferences. Their intake will be weighted using an electronic food scale by a member of the investigation team and then analysed using a nutritional software.

SECONDARY OUTCOMES:
Hunger feelings | immediately after breakfast/lunch/dinner on day 1
  hunger area under the curve will be assessed using visual analogue scale through a the day
Food reward | it will be assessed at dinner baseline
  : The participants will be asked to complete a validated computer-based procedure to measure food reward (Leeds Food Preference Questionnaire; LFPQ). Briefly, the LFPQ provides measures of the wanting and liking for an array of food images, varying in both fat content and taste.

CONTACTS AND LOCATIONS:
Overall Officials: Yves BOIRIE, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Moore H, Pereira B, Fillon A, Miguet M, Masurier J, Beaulieu K, Finlayson G, Thivel D. The association between obesity severity and food reward in adolescents with obesity: a one-stage individual participant data meta-analysis. Eur J Nutr. 2024 Jun;63(4):1241-1255. doi: 10.1007/s00394-024-03348-4. Epub 2024 Feb 20. PMID 38376518